CLINICAL TRIAL: NCT04513353
Title: New Model of Short-term Rehabilitation Exercise Training Using Digital Healthcare System in Patients With Total Knee Arthroplasty; Randomized Controlled Study
Brief Title: Rehabilitation Exercise Using Digital Healthcare System in Patients With Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Jae-Young Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2005/612-001(2)
Record Dates: First submitted 2020-08-09; First posted 2020-08-14 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Total Knee Arthroplasty; Post-Operative Rehabilitation; Digital Healthcare System

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Healthcare System Rehabilitation (Experimental)
  Interventions: Device: Rehabilitation using Digital Healthcare System (Uincare Homeplus)
- Conventional Rehabilitation (Active Comparator)
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Device: Rehabilitation using Digital Healthcare System (Uincare Homeplus) — Uincare Homeplus is a device using infrared, kinect camera and motion capture technology to track 3D motion of the patients' posture and joint articulations. It also has embedded exercise training software dedicated to total knee arthroplasty post-op rehabilitation at home.
  Home-based self-rehabilitation using brochure for 3 weeks post surgery (same as the active comparator)
  Home-based self-rehabilitation using digital healthcare system(Uincare Homeplus) for 3 to 12 weeks post surgery.
  Other Names: Uincare Homeplus
  Arms: Digital Healthcare System Rehabilitation
Other: Conventional Rehabilitation — Home-based self-rehabilitation using brochure for 12 weeks post surgery.
  Arms: Conventional Rehabilitation

SUMMARY:
The study aims to examine the effect of short-term rehabilitation exercise support using digital healthcare system (Uincare homeplus) in the patients with total knee arthroplasty. The study is a two-arm prospective randomized controlled study comparing the effect of rehabilitation exercise digital healthcare system at home with conventional brochure-based home exercise. Gait speed (4-meter), Pain (using Numerical rating scale), knee joint range of motion (ROM), lower extremities motor power (using Manual muscle test), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Berg Balance Scale (BBS) and quality of life using EQ-5D-5L will be evaluation on enrollment, 3-weeks, 6-weeks, 12-weeks and 24-weeks after enrollment.

DETAILED DESCRIPTION:
Total knee arthroplasty is treatment of choice for knee degenerative arthritis patients who are unresponsive to non-operative management including medications and physical therapies. Total knee arthroplasty is an effective treatment enhancing the joint range of motion as well as reducing pain and correcting deformities which leads to better patient function with better quality of life. Current method of post-operative rehabilitation is home-based self rehabilitation using brochure, combined with one or two times of education at the hospital before discharge. Patients often find difficulty in doing rehabilitation by themselves at home without supervision which resulted in decreased compliance.

With development of technologies using multi-motion sensor and AR(augmented-reality) system, the investigators have developed a digital healthcare system(Uincare Homeplus) which can supplement patients' rehabilitation at home by giving them proper instructions as well as feedback. In this prospective randomized controlled study, the investigators aim to compare the efficacy of the newly-developed digital healthcare system with conventional rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had total knee arthroplasty
* Patient who is discharged to home after surgery

Exclusion Criteria:

* Patient who had previous history of high tibial osteotomy on the affected lower extremities.
* Patient who had history of lower extremities joint revision arthroplasty in the past 6 months.
* Patient who has severe comorbidity that inhibits exercise.
* Patient who has major neurological deficits on the lower extremities.
* Patient who cannot participate in post surgery rehabilitation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline Gait Speed | Enrollment, 3-weeks, 6-weeks, 12-weeks, 24-weeks
  Gait Speed is measured by the time required to walk 4-meters in plain indoor. Shorter time required to complete 4-meter walk means better gait function.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) on the affected knee | Enrollment, 3-weeks, 6-weeks, 12-weeks, 24-weeks
  Evaluation of pain of the affected shoulder using numerical rating scale (0-10, with score 0 indicating no pain). the higher score means worse pain.
Range of Motion (ROM) on the affected knee | Enrollment, 3-weeks, 6-weeks, 12-weeks, 24-weeks
  Evaluation of change of ROM in the affected knee from baseline to 24 weeks
Manual Muscle Test (MMT) on the affected lower extremities | Enrollment, 3-weeks, 6-weeks, 12-weeks, 24-weeks
  Evaluation of change of MMT in the affected lower extremities from baseline to 24 weeks. affected lower extremities MMT scales from 0-25, higher score meaning better outcome.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) on the affected knee | Enrollment, 3-weeks, 6-weeks, 12-weeks, 24-weeks
  The WOMAC is a self-administered questionnaire used in the evaluation of knee osteoarthritis. It is consisted with 24 items divided into 3 subscales; Pain, Stiffness and Physical function. WOMAC score ranges from 0-96 with higher score meaning worse pain, stiffness and function.
Berg Balance Scale (BBS) | Enrollment, 3-weeks, 6-weeks, 12-weeks, 24-weeks
  BBS is a 14-item objective measure that assess static balance and fall risk in adults. BBS score ranges from 0-56, with higher score meaning better balance.
Quality of Life using EQ-5D-5L | Enrollment, 3-weeks, 6-weeks, 12-weeks, 24-weeks
  Evaluation of quality of life using EQ-5D-5L. This scale is numbered from -0.066 to 0.904. Lower value means worse quality of life

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shim GY, Kim EH, Lee SJ, Chang CB, Lee YS, Lee JI, Hwang JH, Lim JY. Postoperative rehabilitation using a digital healthcare system in patients with total knee arthroplasty: a randomized controlled trial. Arch Orthop Trauma Surg. 2023 Oct;143(10):6361-6370. doi: 10.1007/s00402-023-04894-y. Epub 2023 May 2. PMID 37129691